CLINICAL TRIAL: NCT00994266
Title: Efficacy of Diamel in the Treatment of Type 2 Diabetic Patients Receiving Insulin Therapy
Brief Title: Diamel in the Treatment of Type 2 Diabetic Patients Receiving Insulin Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Maria Elena de la Uz Herrera, "Abel Santamaría Cuadrado"General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAT-0912-CU
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Diamel; Dietary supplement
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Diamel
  Interventions: Dietary Supplement: Diamel
- B (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Diamel — Two Diamel tablets (Orally administered) three times a day (just before each meal: breakfast, lunch and dinner), for 24 weeks, in combination with the standard treatment consisting in two daily doses of insulin and proper diet.
  Arms: A
Dietary Supplement: Placebo — Two Placebo tablets (Orally administered) three times a day (just before each meal: breakfast, lunch and dinner), for 24 weeks, in combination with the standard treatment consisting in two daily doses of insulin and proper diet.
  Arms: B

SUMMARY:
The purpose of this study is to assess the efficacy of Diamel (dietary supplement) administration in the treatment of patients with type 2 diabetes receiving insulin therapy. The duration of this double-blind placebo controlled phase 3 clinical trial will be 24 weeks. The estimated number of patients to be recruited and randomized for the study is 116. Daily insulin requirements, blood glucose (fasting and post-prandial) concentrations, glycosylated hemoglobin (HbA1c), triglycerides and cholesterol will be assessed at the beginning and after 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes with insulin therapy regimen of two daily doses.
* Signed informed consent.

Exclusion Criteria:

* Type 1 diabetes.
* Type 2 diabetes with glibenclamide treatment.
* Nephropathy or liver condition diagnosed by clinical and/or biochemical examination.
* Sepsis.
* Pregnancy.
* HbA1c values greater than 10%.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2009-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Difference of insulin daily doses at week 24 and at the beginning of the study | 24 weeks
Difference of glucose concentrations (fasting and post-prandial) at week 24 and at the beginning of the study considering the adjusted insulin doses during treatment | 24 weeks

SECONDARY OUTCOMES:
Occurrence of hypoglycemic episodes during treatment | 24 weeks
Difference of HbA1c concentrations at week 24 and at the beginning of the study | 24 weeks
Difference of triglycerides and cholesterol concentrations at week 24 and at the beginning of the study | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elena de la Uz Herrera, MSC, Principal Investigator — "Abel Santamaría Cuadrado" General Hospital; Arturo Hernández Yero, PhD, Study Director — National Institute of Endocrinology
Locations (1):
- Diabetes Care Center. "Abel Santamaría Cuadrado" General Hospital, Pinar del Río, Provincia de Pinar del Río, Cuba